CLINICAL TRIAL: NCT04604405
Title: Effect of 650nm Low Energy Light on Macular Microcirculation in Myopia Prevention and Control
Brief Title: Effects of 650nm Low Energy Light on Human Retina and Choroid Microcirculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, jun ren, Attending doctor,Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cq-wy-pbm-01
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Myopia
Keywords: photobiomodulation,macular microcirculation,,myopia
MeSH Terms: conditions — Myopia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photobiomodulation (Experimental): Eyes are irradiated with 650nm low energy red light
  Interventions: Radiation: photobiomodulation
- blank (No Intervention): no intervention except for wear glasses

INTERVENTIONS:
Radiation: photobiomodulation — 650nm low energy red light eye irradiation
  Arms: photobiomodulation

SUMMARY:
This project is a single-center, prospective, self-controlled clinical study. It intends to select patients with simple medium and low degree myopia as subjects, and apply 650nm low-energy red light irradiation to the retina to observe its effect on macular microcirculation.

DETAILED DESCRIPTION:
A total of 120 subjects are planned to be recruited and divided into 4 groups according to age and intervention, including 30 in the juvenile intervention group, 30 in the juvenile control group, 30 in the adult intervention group and 30 in the adult control group. Two intervention groups received 650nm low-energy red light irradiation treatment with a 650nm low-energy light emitter, twice a day for 3 minutes each time, The subjects were treated and followed up for 3 months. The control group was not treated and followed up for 3 months too. All subjects were followed up before treatment, at the end of the 1st month and at the end of 3rd month. Angio-oct was used as the main examination to observe and record the vascular density and blood perfusion in macular area. Axial length, diopter and OCT were used as secondary observation indexes. At the end of the experiment, the data of the intervention group and the control group were compared

ELIGIBILITY:
Inclusion Criteria:

1. Age from 7 to 17 years old or from 18 to 45 years old;
2. Meet the diagnostic criteria for patients with simple low or moderate myopia, with diopter < -6.0d and eye axis < 26.0mm;
3. Transparent refractive stroma, no other eye diseases except nearsightedness;
4. Agree to participate in the clinical study and sign the informed consent.

Exclusion Criteria:

1. Other ocular lesions, such as uveitis, retinal/choroidal vascular lesions, congenital ocular lesions, glaucoma, high myopia (ocular axis > 26cm), degenerative retinal disease, optic neuropathy, etc.;
2. Another eye with low vision
3. Corneal edema/epithelial detachment, corneal opacity;
4. Redness, pain, dry eye, photophobia, difficulty in opening eyes;
5. Had a history of eye surgery in recent 3 months;
6. Severe impairment of liver and kidney function and/or serious systemic diseases (such as cardiovascular, respiratory, digestive, nervous, endocrine, genitourinary, etc.);
7. Women who are already pregnant, preparing for pregnancy during the study period and lactating;
8. A history of substance abuse or alcohol abuse;
9. Receiving prevention and control treatment for myopia other than glasses within the first 30 days;
10. Any situation in which the study physician believes that the patient's condition will interfere with the clinical study (e.g., the patient is prone to nervous tension, uncontrollable emotions, depression, etc.)

Ages: 7 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
retinal vascular density | 12 weeks
  The vascular density of the inner retinal layer in the macular area within 3×3mm was measured by angio-OCT
retinal vascular perfusion | 12 weeks
  The perfusion of the inner retinal layer in the macular area within 3×3mm was measured by angio-OCT
Choroid thickness | 12 weeks
  Distance from Bruch membrane to The inner surface of the sclera

SECONDARY OUTCOMES:
Axial length | 12 weeks
  Distance from corneal apex to macular fovea
diopter | 12 weeks
  Myopic degree

CONTACTS AND LOCATIONS:
Overall Officials: yi wang, master, Study Director — Doctoral supervisor
Locations (1):
- Chongqing Aier Eye Hosipital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ren J, Xu JN, Liu YZ, Gu XL, Wang Y. Short-term effectiveness and safety of photobiomodulation on low-to-moderate myopia. Lasers Med Sci. 2025 Feb 15;40(1):95. doi: 10.1007/s10103-024-04119-7. PMID 39954097